CLINICAL TRIAL: NCT02293850
Title: A Phase I Study to Evaluate the Safety and Efficacy of Telomelysin (OBP-301) in Patients With Hepatocellular Carcinoma
Brief Title: Phase I Study to Evaluate the Safety and Efficacy of Telomelysin (OBP-301) in Patients With Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oncolys BioPharma Inc (Industry)
Collaborators: Medigen Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-OT-21
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single intra-tumoral injection (Experimental): OBP-301 ; Cohort 1: 1x10 10 viral particle (VP)/ tumor Cohort 2: 1x10 11 viral particle (VP)/ tumor Cohort 3: 1x10 12 viral particle (VP)/ tumor
  Interventions: Biological: OBP-301

INTERVENTIONS:
Biological: OBP-301 — A range of dose levels is investigated and the starting dose is 1x1010 VP/tumor. Dose administration will be conducted through a dose-escalating scheme from 1x1010 VP/tumor to 1x1011 VP/tumor, 1x1012 VP/tumor, 3x1011 VP/tumor and 3x1012 VP/tumor.

SUMMARY:
This is an open labeled, multiple centers, two countries (Taiwan and Korea) non-comparative phase I trial in patients with hepatocellular carcinoma. In phase I part, a maximum of 18 patients will be recruited in this study.

DETAILED DESCRIPTION:
After screening, each eligible patient will undergo a treatment of OBP-301 within 14 days and will automatically enter follow-up period.

The follow-up period is up to 12 weeks after the last injection in the phase I part.

Each patient will return for follow-up visit weekly in the first month after the last injection, and then every 4 weeks up to the end of follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 65 years (19 to 65 years in Korea), either sex
2. Patients diagnosed with hepatocellular carcinoma. The diagnosis of HCC (hepatocellular carcinoma) should be established by cytology or histopathology
3. Patients who have unresectable HCC and meet all of the following conditions:

   * Barcelona Clinic Liver Cancer (BCLC) stage B or C
   * TransAarterial ChemoEmbolization (TACE) refractory in discretion of the investigators, or TACE unsuitable (such as but not limited to portal vein thrombosis)
   * Local ablative treatment (such as percutaneous ethanol injection, radiofrequency ablation, etc) unsuitable
   * Sorafenib failure, intolerable or ineligible
4. Patients must have at least one lesion that can be accurately measured in at least one dimension as 1 cm or more and the lesion must be suitable for repeat measurement
5. Patients who have Child-Pugh's Score no greater than 7, and have no ascites
6. Patients who have all the conditions below at screening:

   serum ALT (Alanine Aminotransferase) level (GPT) less than 2.5 x UNL
   * serum AST (Aspartate Aminotransferase) level (GOT) less than 2.5 x UNL
   * WBC (white blood cell) greater than or equal to 3,000 / microliter
   * Serum creatinine less than or equal to 1.5 x UNL
   * activated partial thromboplastin time (APTT) <1.5 x UNL
7. Platelet count correctable to greater than or equal to 80,000 / microliter
8. prothrombin time-international normalized ratio (PT-INR) correctable to less than 1.5
9. Patients who have life expectancy longer than 12 weeks

Exclusion Criteria:

1. Patients who have had chemotherapy within last three weeks (6 weeks for nitrosourea or Mitomycin-C) prior to dosing
2. Patients who have had radiotherapy to tumor site within the last four weeks prior to dosing and with documentation of subsequent tumor growth at this site
3. Patients who have received other investigational or antineoplastic medication within the last four weeks prior to dosing
4. Patients who had history of esophageal variceal bleeding within eight weeks prior to study entry
5. Patients who have uncontrolled diabetes, active or chronic infection, including HIV, except for asymptomatic bacterial colonization, hepatitis B virus (HBV), or hepatitis C virus (HCV) infection
6. Patients who had acute viral infection syndrome diagnosed within the last two weeks
7. Patients who have concomitant hematological malignancy (e.g. acute lymphocytic leukemia, non-Hodgkin's lymphoma)
8. Patients who have active rheumatoid arthritis or other autoimmune disease.
9. Patients who have current requirement for chronic systemic immunosuppressive medication including any dose of glucocorticoid or cyclosporin, or chronic use of any such medication within the last four weeks Note: Course of glucocorticoid therapy less than 10 days duration is allowed (e.g. for nausea control)
10. Patients with organ transplants (may require prolonged immunosuppressive therapy)
11. Patients who had prior participation in any research protocol which involved administration of adenovirus vectors
12. Patients received any immune-related related related related related blood products, such as immunoglobulin in the prior 3 months
13. Patients who have uncontrolled concurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
14. Psychiatric, addictive, or any disorder which compromises ability to give truly informed consent for participation in this study or adequate compliance
15. Female patients that are pregnant or on breast-feeding
16. Patients who receive anti-platelet agents or anti-coagulation agents (e.g. Heparin, warfarin, aspirin, ticlopidine, clopidogrel, dipyridamole and so on).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of safety parameters (adverse events, laboratory data, EKG, body weight, vital signs) on patient-base. | 14 weeks

SECONDARY OUTCOMES:
Maximum Tolerated Dose (MTD)/ Maximum Feasible Dose (MFD) for patients using OBP-301. | 16 weeks
Dose-Limiting Toxicity (DLT) for patients using OBP-301. | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jer Chen, M.D., Ph.D., Study Chair — National Taiwan University Hospital
Locations (2):
- Pusan National University Hospital, Busan, South Korea
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Heo J, Liang JD, Kim CW, Woo HY, Shih IL, Su TH, Lin ZZ, Yoo SY, Chang S, Urata Y, Chen PJ. Safety and dose escalation of the targeted oncolytic adenovirus OBP-301 for refractory advanced liver cancer: Phase I clinical trial. Mol Ther. 2023 Jul 5;31(7):2077-2088. doi: 10.1016/j.ymthe.2023.04.006. Epub 2023 Apr 14. PMID 37060176